CLINICAL TRIAL: NCT01594970
Title: A Safety and Efficacy Study of Bimatoprost 0.01% in Primary Open-Angle Glaucoma (POAG) or Ocular Hypertension (OH)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: APMA-001211
Record Dates: First submitted 2012-05-08; First posted 2012-05-09 (Estimated); Results first posted 2014-01-28 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bimatoprost 0.01% (Naive Monotherapy) (Experimental): 1 drop in the affected eye(s), administered in the evening in previously treatment naive subjects for 12 weeks.
  Interventions: Drug: Bimatoprost 0.01%
- Bimatoprost 0.01% (Switched Monotherapy) (Experimental): 1 drop in the affected eye(s), administered in the evening in subjects who were previously on another monotherapy treatment for 12 weeks.
  Interventions: Drug: Bimatoprost 0.01%
- Bimatoprost 0.01% (with Adjunctive Therapy) (Experimental): 1 drop in the affected eye(s), administered in the evening in subjects who are also receiving adjunctive therapy for 12 weeks.
  Interventions: Drug: Bimatoprost 0.01%

INTERVENTIONS:
Drug: Bimatoprost 0.01% — 1 drop in the affected eye(s), administered in the evening for 12 weeks.
  Other Names: LUMIGAN® 0.01%

SUMMARY:
This study will evaluate the safety and efficacy of bimatoprost 0.01% in subjects with elevated intraocular pressure (IOP) due to primary open-angle glaucoma (POAG) or ocular hypertension (OH).

ELIGIBILITY:
Inclusion Criteria:

* Elevated IOP due to either primary open-angle glaucoma or ocular hypertension

Exclusion Criteria:

* None

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2012-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Seoul, South Korea

REFERENCES:
- [Derived] Park KH, Simonyi S, Kim CY, Sohn YH, Kook MS. Bimatoprost 0.01% in treatment-naive patients with open-angle glaucoma or ocular hypertension: an observational study in the Korean clinical setting. BMC Ophthalmol. 2014 Dec 17;14:160. doi: 10.1186/1471-2415-14-160. PMID 25519810

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bimatoprost 0.01% (Naive Monotherapy) | Bimatoprost 0.01% (Switched Monotherapy) | Bimatoprost 0.01% (With Adjunctive Therapy)
Started | 295 | 248 | 257
Completed | 220 | 166 | 191
Not Completed | 75 | 82 | 66
Not completed — Non-Adverse Event Related | 4 | 5 | 6
Not completed — Adverse Event | 17 | 23 | 23
Not completed — Lost to Follow-up | 54 | 54 | 37

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimatoprost 0.01% (Naive Monotherapy) | Bimatoprost 0.01% (Switched Monotherapy) | Bimatoprost 0.01% (With Adjunctive Therapy) | Total
Number analyzed (Participants) | 295 | 248 | 257 | 800
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.0 (13.81) | 59.5 (13.23) | 61.2 (12.59) | 59.5 (13.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 145 | 105 | 380
  Male | 165 | 103 | 152 | 420

OUTCOME MEASURES:

1. Primary Outcome: Severity of Ocular Hyperemia in the Study Eye on a 5-Point Scale
Description: Hyperemia is the engorgement of the blood vessels (redness) of the eye. Hyperemia is graded in the study eye on a 5 point scale where 0=None (Normal), 0.5=Trace (Trace reddish pink with no more than slight perilimbal injection), 1=Mild (Mild flush reddish color), 2=Moderate (Bright red color), and 3=Severe (Deep, bright, diffuse redness). The numbers of participants in each severity grade are presented.
Time Frame: Week 12
Population: Intent to Treat: all treated subjects with data at this time point
Measure: Number; unit: Participants
Arm/Group | Bimatoprost 0.01% (Naive Monotherapy) | Bimatoprost 0.01% (Switched Monotherapy) | Bimatoprost 0.01% (With Adjunctive Therapy)
Number analyzed (Participants) | 220 | 166 | 191
Participants
  None | 40 | 49 | 20
  Trace | 71 | 54 | 70
  Mild | 73 | 47 | 65
  Moderate | 31 | 11 | 30
  Severe | 5 | 5 | 6

2. Secondary Outcome: Change From Baseline in Intraocular Pressure (IOP)
Description: IOP is a measure of the fluid pressure inside the eye. A negative number change from baseline indicates a reduction in IOP (improvement).
Time Frame: Baseline, Week 6, Week 12
Population: Intent to Treat: all treated subjects
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Bimatoprost 0.01% (Naive Monotherapy) | Bimatoprost 0.01% (Switched Monotherapy) | Bimatoprost 0.01% (With Adjunctive Therapy)
Number analyzed (Participants) | 295 | 248 | 257
Millimeters of Mercury (mmHg)
  Baseline | 18.6 (5.39) | 17.0 (5.73) | 19.3 (6.19)
  Change from Baseline at Week 6 (N=251, 204, 233) | -4.7 (4.50) | -2.6 (4.43) | -3.2 (5.44)
  Change from Baseline at Week 12 (N=220, 165, 191) | -4.3 (4.42) | -2.8 (4.68) | -3.4 (6.11)

3. Secondary Outcome: Overall Percent Change From Baseline in IOP
Description: IOP is a measure of the fluid pressure inside the eye. A negative number change response indicates a reduction in IOP (improvement).
Time Frame: Baseline, Week 6, Week 12
Population: Intent to Treat: all treated subjects with data at this time point
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Bimatoprost 0.01% (Naive Monotherapy) | Bimatoprost 0.01% (Switched Monotherapy) | Bimatoprost 0.01% (With Adjunctive Therapy)
Number analyzed (Participants) | 295 | 248 | 257
Percent Change
  Change from Baseline at Week 6 (N=251, 204, 233) | -22.09 (17.023) | -12.90 (18.912) | -14.37 (20.883)
  Change from Baseline at Week 12 (N=220, 165, 191) | -20.22 (17.566) | -12.81 (19.438) | -14.25 (23.376)

4. Other Pre Specified Outcome: Change From Baseline in Hyperemia Severity in the Study Eye
Description: Hyperemia is the engorgement of the blood vessels (redness) of the eye. Hyperemia was graded in the study eye on a 5 point scale where 0=None (Normal), 0.5=Trace (Trace reddish pink with no more than slight perilimbal injection), 1=Mild (Mild flush reddish color), 2=Moderate (Bright red color), and 3=Severe (Deep, bright, diffuse redness). 'Lower' categories refer to grades 0, 0.5 and 1, and 'higher' categories refer to grades 2 and 3. Change in hyperemia severity was classified as improved, no change or worsened based on the change in the hyperemia grading category from higher to lower, no change in category or lower to higher, respectively. The numbers of participants in each category are presented.
Time Frame: Baseline, Week 12
Population: Intent to Treat: all treated subjects with data at this time point
Measure: Number; unit: Participants
Arm/Group | Bimatoprost 0.01% (Naive Monotherapy) | Bimatoprost 0.01% (Switched Monotherapy) | Bimatoprost 0.01% (With Adjunctive Therapy)
Number analyzed (Participants) | 220 | 166 | 191
Participants
  Improved | 1 | 8 | 15
  No Change | 191 | 149 | 159
  Worsened | 28 | 9 | 17

ADVERSE EVENTS:
Arm/Group | Bimatoprost 0.01% (Naive Monotherapy) | Bimatoprost 0.01% (Switched Monotherapy) | Bimatoprost 0.01% (With Adjunctive Therapy)
Serious Adverse Events (participants affected / at risk) | 1/295 | 0/248 | 1/257
Other Adverse Events (participants affected / at risk) | 7/295 | 9/248 | 14/257
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost 0.01% (Naive Monotherapy) (N=295) | Bimatoprost 0.01% (Switched Monotherapy) (N=248) | Bimatoprost 0.01% (With Adjunctive Therapy) (N=257)
Glaucoma (Eye disorders) | 0 | 0 | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost 0.01% (Naive Monotherapy) (N=295) | Bimatoprost 0.01% (Switched Monotherapy) (N=248) | Bimatoprost 0.01% (With Adjunctive Therapy) (N=257)
Conjunctival Hyperaemia (Eye disorders) | 7 | 9 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is at least 30 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.